CLINICAL TRIAL: NCT01628640
Title: Phase I Trial of Intratumoral Injection of Vesicular Stomatitis Virus Expressing Human Interferon Beta in Patients With Sorafenib Refractory/Intolerant Hepatocellular Carcinoma, Advanced Solid Tumors With Liver Predominant Locally Advanced/Metastatic Disease or Subcutaneous/Cutaneous Lesions
Brief Title: Viral Therapy in Treating Patient With Refractory Liver Cancer or Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1148; NCI-2012-00890 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 11-007114 (Other: Mayo Clinic Institutional Review Board); MC1148 (Other: Mayo Clinic); 4781 (Other Grant/Funding Number: OPD Grant); P50CA210964 (NIH); R01FD004781 (FDA); DP2CA195764 (NIH)
Record Dates: First submitted 2012-06-23; First posted 2012-06-27 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Advanced Malignant Solid Neoplasm; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (viral therapy in single tumor location) (Experimental): Patients with hepatocellular carcinoma or advanced solid tumor with liver lesions receive recombinant vesicular stomatitis virus expressing interferon beta intratumorally in a single tumor location on day 1.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Biological: Recombinant Vesicular Stomatitis Virus-expressing Interferon-beta
- Arm B (viral therapy in multiple locations) (Experimental): Patients with advanced solid tumor with subcutaneous/cutaneous lesions receive recombinant vesicular stomatitis virus expressing interferon beta intratumorally in up to 5 cutaneous, subcutaneous, or soft tissue tumor lesions on day 1.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Biological: Recombinant Vesicular Stomatitis Virus-expressing Interferon-beta

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Biological: Recombinant Vesicular Stomatitis Virus-expressing Interferon-beta — Given intratumorally
  Other Names: Recombinant VSV-IFN-beta; VSV-hIFN-b

SUMMARY:
This phase I trial studies the best dose and side effects of recombinant vesicular stomatitis virus expressing interferon beta in treating patients with liver cancer or solid tumors with lesions that have spread to other parts of the body and do not respond to treatment. The study virus has a gene inserted into it which will allow production of interferon beta, which is a substance that will restrict the spread of the virus to tumor cells and not healthy cells. It will also have some independent anti-cancer activity. Although the primary goal of this study is to evaluate the safety of delivery of this viral agent to people, patients may benefit clinically by having shrinkage or stabilization of their tumor or reduction in their cancer related symptoms (e.g., pain). Funding Source - FDA OOPD.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of recombinant vesicular stomatitis virus-expressing interferon-beta (VSV-IFN-beta) in patients with hepatocellular carcinoma (HCC) refractory or intolerant to sorafenib therapy and patients with advanced solid tumors with liver predominant locally advanced/metastatic treatment refractory disease. (Arm A) II. To determine the maximum tolerated dose (MTD) of VSV-IFN-beta in patients with advanced solid tumors with subcutaneous/cutaneous lesions. (Arm B)

SECONDARY OBJECTIVES:

I. To estimate the tumor response rate, injected lesion (TNi) and distant lesion (TNd) necrosis rate (with TNi and TNd response defined as >= 30% increase in necrosis from baseline) and overall survival. (Arm A)

TERTIARY OBJECTIVES:

I. To determine the pharmacokinetic (PK) profile of VSV-IFN-beta in patients with HCC by or advanced solid tumors with liver predominant disease or subcutaneous/cutaneous lesions by measurement of VSV-IFN-beta in blood by reverse transcriptase polymerase chain reaction (RT-PCR).

II. To characterize the pharmacodynamics (PD) of VSV-IFN-beta by way of measuring serum interferon-beta and also VSV-RT-PCR of VSV-IFN-beta listed above.

III. Assess CD8+ T cell (both general and VSV-hIFN-beta specific) and natural killer (NK) cell responses.

IV. Assess status of human interferon beta pathway pre/post therapy in tumor/normal liver tissue (status of IFN-beta, interferon stimulated gene factor 3 [ISGF3 complex constituting signal transducer and activator of transcription (STAT)1/2 and p48 (ISGF3 gamma)]).

V. Assess phosphorylation of STAT1/2 post-therapy. VI. Evaluate transcription of interferon mediated genes (protein kinase R, the death receptor-tumor necrosis factor [TNF]-related apoptosis-inducing ligand [TRAIL], 2'-5' oligoadenylate/ribonucleic acid [RNA]se L proteins, heat shock proteins [Hsp 60/70/90], major histocompatibility class antigens and interferon regulatory factor [IRF]-7).

VII. Assess presence of VSV in tumor/normal liver subsequent to administration of VSV-human IFN-beta (hIFN- beta).

VIII. For HCC patients only, assess preliminary relationships between hepatitis C genotype (in those patients that are hepatitis C positive) and any evidence of anti-tumor efficacy.

OUTLINE: This is a dose-escalation study. Patients are assigned to 1 of 2 arms.

ARM A: Patients with hepatocellular carcinoma or advanced solid tumor with liver lesions receive recombinant vesicular stomatitis virus expressing interferon beta intratumorally in a single tumor location on day 1.

ARM B: Patients with advanced solid tumor with subcutaneous/cutaneous lesions receive recombinant vesicular stomatitis virus expressing interferon beta intratumorally in up to 5 lesions on day 1.

After completion of study treatment, patients are followed up every 4 weeks for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* ARM A: Histologically or cytologically confirmed hepatocellular carcinoma that is refractory (by Response Evaluation Criteria in Solid Tumors [RECIST] or modified [m]RECIST criteria or with unequivocal clinical progression of disease) to or intolerant (defined as inability to administer further sorafenib due to drug related toxicities) of sorafenib based therapy or advanced solid tumor with liver predominant disease burden that has progressed on or is intolerant to standard
* ARM A: Absolute neutrophil count (ANC) >= 1000/mm^3
* ARM A: Platelet count >= 80,000/mm^3
* ARM A: Hemoglobin >= 10 g/dl
* ARM A: Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 5 x ULN
* ARM A: Creatinine =< 1.5 x ULN
* ARM A: Total bilirubin =< 1.5 x ULN
* ARM A: International normalized ratio (INR) =< 1.5 x ULN
* ARM A: Activated partial thromboplastin time (aPTT) =< 1.5 x ULN
* ARM A: Ability to provide informed written consent
* ARM A: Willingness to return to Mayo Clinic in Arizona for follow-up
* ARM A: Life expectancy >= 12 weeks
* ARM A: Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* ARM A: Willingness to provide all biological specimens as required by the protocol
* ARM A: Negative serum pregnancy test =< 7 days prior to registration for women of childbearing potential only
* ARM A: Child Pugh Score A or B7 (patients with ascites must have paracentesis performed within scope of standard of care, to be able to successfully perform intratumoral injection procedure)
* ARM A: The patient and their partner agree to use a barrier method of contraception during the study and 4 months following end of active treatment
* ARM A: Disease burden in liver not affecting more than 25% of liver
* ARM A: Predominant intrahepatic burden (> 75%) of disease (i.e. patients with widespread extrahepatic disease to organs other than the liver will not be included)
* ARM B: Histologically or cytologically confirmed solid tumor with subcutaneous/cutaneous lesions that is refractory (RECIST or with unequivocal clinical progression of disease) to or intolerant to standard therapy
* ARM B: Absolute neutrophil count (ANC) >= 1000/mm^3
* ARM B: Platelet count >= 100,000/mm^3
* ARM B: Hemoglobin >= 10 g/dl
* ARM B: AST/ALT =< 2.5 x ULN
* ARM B: Creatinine =< 1.5 x ULN
* ARM B: Total bilirubin =< 1.5 x ULN
* ARM B: INR =< 1.5 x ULN
* ARM B: aPTT =< 1.5 x ULN
* ARM B: Ability to provide informed written consent
* ARM B: Willingness to return to Mayo Clinic in Arizona for follow-up
* ARM B: Life expectancy >= 12 weeks
* ARM B: ECOG performance status (PS) 0 or 1
* ARM B: Willingness to provide all biological specimens as required by the protocol
* ARM B: Negative serum pregnancy test =< 7 days prior to registration for women of childbearing potential only
* ARM B: Child Pugh Score A
* ARM B: The patient and their partner agree to use a barrier method of contraception during the study and 4 months following end of active treatment
* ARM B: Disease burden in liver not affecting more than 25% of liver

Exclusion Criteria:

* ARM A: Uncontrolled infection
* ARM A: Systemic anti-cancer therapy =< 4 weeks prior to registration
* ARM A: Known human immunodeficiency virus (HIV) infection
* ARM A: Other concurrent chemotherapy, immunotherapy, radiotherapy, or investigational therapy
* ARM A: Pregnant or nursing women
* ARM A: History of bone marrow or solid organ transplantation
* ARM A: Patient for whom surgical resection or liver transplantation would be more appropriate
* ARM A: Any condition, which in the opinion of the investigator would render the patient unsuitable to participate in the study
* ARM A: Any corticosteroid use =< 28 days prior to registration
* ARM A: Any radioembolization or transarterial chemoembolization (TACE) =< 84 days prior to registration
* ARM B: Uncontrolled infection
* ARM B: Systemic anti-cancer therapy =< 4 weeks prior to registration
* ARM B: Known HIV infection
* ARM B: Other concurrent chemotherapy, immunotherapy, radiotherapy, or investigational therapy
* ARM B: Pregnant or nursing women
* ARM B: History of bone marrow or solid organ transplantation
* ARM B: Patient for whom surgical resection or liver transplantation would be more appropriate
* ARM B: Any condition, which in the opinion of the investigator would render the patient unsuitable to participate in the study
* ARM B: Any corticosteroid use =< 28 days prior to registration
* ARM B: Any radioembolization or TACE =< 84 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-08-03 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-04-19 (Actual)

PRIMARY OUTCOMES:
Best tumor response, defined as the best objective status recorded among patients with measurable disease at baseline using Response Evaluation Criteria in Solid Tumors version 1.1 | From the start of the treatment until disease progression, assessed up to 3 years
  Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease in this patient population (overall, by dose level, and by disease type). Examined in an exploratory and hypothesis-generating fashion.
Incidence of adverse events, graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 3 years
  All eligible patients that have initiated treatment will be considered evaluable for assessing adverse event rate(s). The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed by dose level to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration. Examined in an exploratory and hypothesis-generating fashion.
Maximum tolerated dose, defined as the highest dose at which no more than 1/6 patients experiences dose limiting toxicities, graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | 4 weeks
  Dose limiting toxicities defined as an adverse event during the first 4 weeks following injection. A modified "3+3" Fibonacci dose escalation scheme will be used Examined in an exploratory and hypothesis-generating fashion.
Overall survival | From registration to death due to any cause, assessed up to 3 years
  The distribution of survival time will be estimated using the method of Kaplan-Meier (overall, by dose level, and by disease type). Examined in an exploratory and hypothesis-generating fashion.
Tumor necrosis | Up to 3 years
  Injected lesion and distant lesion necrosis rate will be defined as injected lesion and distant lesion >= 30% increase in necrosis from baseline, respectively. Frequency and relative frequency will be computed for each (overall, by dose level and by disease type). This analysis will be conducted in hepatocellular carcinoma patients only.

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh J. Borad, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- [Derived] Nagalo BM, Zhou Y, Loeuillard EJ, Dumbauld C, Barro O, Elliott NM, Baker AT, Arora M, Bogenberger JM, Meurice N, Petit J, Uson PLS Jr, Aslam F, Raupach E, Gabere M, Basnakian A, Simoes CC, Cannon MJ, Post SR, Buetow K, Chamcheu JC, Barrett MT, Duda DG, Jacobs B, Vile R, Barry MA, Roberts LR, Ilyas S, Borad MJ. Characterization of Morreton virus as an oncolytic virotherapy platform for liver cancers. Hepatology. 2023 Jun 1;77(6):1943-1957. doi: 10.1002/hep.32769. Epub 2022 Oct 11. PMID 36052732
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials